CLINICAL TRIAL: NCT03832816
Title: Behavioral and Physiological Effects of delta9-Tetrahydrocannabinol (THC) and Cannabidiol (CBD)
Brief Title: Behavioral and Physiological Effects of THC and CBD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: cancellation of funding contract
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00199386
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers
Keywords: cortisol; ACTH; Heart rate; delta9-Tetrahydrocannabinol; cannabidiol
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): Distilled Water
  Interventions: Drug: Placebo
- Vaporized THC alone (Experimental): 5mg pure THC
  Interventions: Drug: Vaporized THC alone
- Vaporized low CBD alone (Experimental): 50mg pure CBD
  Interventions: Drug: Vaporized CBD alone
- Vaporized medium CBD alone (Experimental): 100mg pure CBD
  Interventions: Drug: Vaporized CBD alone
- Vaporized high CBD alone (Experimental): 200mg pure CBD
  Interventions: Drug: Vaporized CBD alone
- Vaporized low CBD with THC (Experimental): 50mg pure CBD paired with 5mg THC
  Interventions: Drug: Vaporized CBD with THC
- Vaporized medium CBD with THC (Experimental): 100mg pure CBD paired with 5mg THC
  Interventions: Drug: Vaporized CBD with THC
- Vaporized high CBD with THC (Experimental): 200mg pure CBD paired with 5mg THC
  Interventions: Drug: Vaporized CBD with THC

INTERVENTIONS:
Drug: Placebo — Placebo vapor (distilled water)
  Other Names: distilled water
  Arms: Placebo
Drug: Vaporized THC alone — Acute exposure to vaporized THC
  Arms: Vaporized THC alone
Drug: Vaporized CBD alone — Acute exposure to vaporized CBD
  Arms: Vaporized high CBD alone; Vaporized low CBD alone; Vaporized medium CBD alone
Drug: Vaporized CBD with THC — Acute exposure to vaporized CBD with THC
  Arms: Vaporized high CBD with THC; Vaporized low CBD with THC; Vaporized medium CBD with THC

SUMMARY:
This study will evaluate physiological and behavioral responses to vaporized delta9-Tetrahydrocannabinol (THC) and cannabidiol (CBD) administered via inhalation.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). In this between-subjects study, participants will be randomized to complete 1 of 8 possible acute drug administration sessions in which participants will administer THC alone, CBD alone, THC and CBD together, or placebo. Following drug administration, participants will complete a performance session and complete a battery of questionnaires assessing subjective drug effects, mood, affect, and mental state. Vital signs and hormone levels will also be assessed before and after drug administration. The study will help the investigators understand the individual and interactive effects of THC and CBD, the two most common cannabis constituents.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent
* Be between the ages of 18 and 50
* Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
* Willingness to provide urine sample at the screening visit and again upon admission for the experimental session
* Test negative for recent drug or alcohol use at the screening visit and upon arrival for each experimental session.
* Not be pregnant or nursing (if female). All females must have a negative pregnancy test at the screening visit and at clinic admission.
* BMI 18-36
* Blood pressure at screening visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Occasional/Intermittent cannabis users.
* Have not donated blood in the prior 30 days.

Exclusion Criteria:

* Recent non-medical use of psychoactive drugs;
* History of or current evidence of significant medical or psychiatric illness
* any condition (as determined by the study physician or investigator) that puts the participant at greater risk.
* Recent use of an over the counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Recent use of a prescription medication (with the exception of hormonal birth control prescriptions) which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject. This includes any medication metabolized via CYP2D6, CYP2C9, CYP2B10, or which induce/inhibit CYP3A4 enzymes.
* Recent use of hemp seeds or hemp oil.
* Recent use of dronabinol (Marinol).
* History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
* Recently enrolled in another clinical trial or have recently received any drug as part of a research study.
* Epilepsy or a history of seizures.
* Individuals who have a recent history of traumatic brain injury diagnosed by CT/MRI and have current sequela from prior brain injury, as determined by the study physician
* Individuals with anemia
* 5th grade reading level or lower.
* Clinically relevant anxiety.
* Individuals who are night shift workers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood cortisol levels | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in blood cortisol levels in micrograms per deciliter (ug/dl) will be measured
Change in blood Adrenocorticotropic hormone (ACTH) levels | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in blood ACTH levels in picograms per milliliter (pg/ml) will be measured
Change in heart rate | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in rate (in beats per minute)
Change in State Anxiety levels as assessed by the State-Trait Anxiety Inventory (STAI) | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in composite STAI score. Scale consists of 20 items assessing state anxiety levels; each item is on 4 point Likert scale ranging from 1 (not at all) to 4 (almost always). Items are summed to obtain a composite score which can range from 20 to 80 (higher scores indicate more anxiety).
Change in Mood state as assessed by the The Profile of Mood States (POMS) | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in total tension-anxiety sub-scale score for POMS. This sub-scale of the POMS consists of 9 items, each on a 4-point Likert scale ranging from 1 (not at all) to 4 (extremely) which are summed to create a total score of 9 to 36 (higher scores indicate more tension/anxiety).
Change in Positive affect levels as assessed by The Positive and Negative Affect Schedule (PANAS) | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in total positive affect score. This PANAS consists of 20 items assessing positive affect (10 items) and negative affect (10 items). Each item is on a 5-point Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely). 10 positive affect items are summed to create a total positive affect score while the 10 negative affect items are summed to create a total negative affect score; higher total scores indicate more positive affect or more negative (i.e., worse) affect.
Change in Negative affect levels as assessed by The Positive and Negative Affect Schedule (PANAS) | Prior to drug exposure and for 4 hours post-exposure.
  Peak change in total negative affect score. This PANAS consists of 20 items assessing positive affect (10 items) and negative affect (10 items). Each item is on a 5-point Likert scale ranging from 1 (very slightly or not at all) to 5 (extremely). 10 positive affect items are summed to create a total positive affect score while the 10 negative affect items are summed to create a total negative affect score; higher total scores indicate more positive affect or more negative (i.e., worse) affect.
Subjective rating of "Drug Effect" as assessed via the Drug Effect Questionnaire | Prior to drug exposure and for 4 hours post-exposure.
  Visual Analog Scale rating of subjective drug effect. Score ranges from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Weerts, PhD, Principal Investigator — Johns Hopkins University; Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States